CLINICAL TRIAL: NCT03469947
Title: Tranexamic Acid in Prehospital and In Hospital Civilian Trauma Care in Antifibrinolytic Therapy Study
Brief Title: California Prehospital and In Hospital Antifibrinolytic Therapy Via TXA
Acronym: Cal-PAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Principal Investigator, Michael Neeki, Director of Research - Emergency Medicine, Arrowhead Regional Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001
Record Dates: First submitted 2018-03-08; First posted 2018-03-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Hemorrhagic Shock; Trauma Injury
Keywords: Tranexamic Acid; TXA
MeSH Terms: conditions — Shock, Hemorrhagic; Accidental Injuries | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Prospective observational cohort administered TXA prehospital and a retrospective cohort for matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prehospital Tranexamic Acid (Experimental): 1 gram of Tranexamic Acid will be given during medical transport
  Interventions: Drug: Tranexamic Acid
- Matched Controls (No Intervention): Retrospective matched controls

INTERVENTIONS:
Drug: Tranexamic Acid — 1 gram of prehospital Tranexamic Acid
  Arms: Prehospital Tranexamic Acid

SUMMARY:
The California Prehospital Antifibrinolytic Therapy (Cal-PAT) study seeks to evaluate the safety and efficacy of Tranexamic Acid (TXA) use in the civilian prehospital and in hospital setting in cases of traumatic hemorrhagic shock.

DETAILED DESCRIPTION:
The Cal-PAT study is a multi-centered, prospective, observational cohort study. From March 2015 to July 2017, patients ≥ 18-years-old who sustained blunt or penetrating trauma with signs of hemorrhagic shock identified were considered for TXA treatment by first responders in the prehospital setting and physicians in hospital. A control group was formed of patients seen in the five years prior to data collection cessation (June 2012 to July 2017) at each receiving center who were not administered TXA. Control group patients were selected through propensity score matching based on gender, age, injury severity scores, and mechanism of injury. The primary outcome measured was mortality. Secondary outcomes measured included the total blood products transfused, the hospital and intensive care unit length of stay, and the incidence of known adverse events associated with TXA.

ELIGIBILITY:
Inclusion Criteria:

* Blunt or penetrating trauma with signs and symptoms of hemorrhagic shock
* Systolic blood pressure less than 90 mmHg at scene of injury, during air and/or ground medical transport, or on arrival to designated trauma centers
* Any sustained blunt or penetrating injury within 3 hours
* Patient who are considered to be at high risk for significant hemorrhage

  1. Estimated blood loss of 500 milliliters int he field accompanied with HR >120
  2. Bleeding not controlled by direct pressure or tourniquet
  3. Major amputation of any extremity above the wrists and above the ankles

Exclusion Criteria:

* Any patient under 18 years of age
* Any patient with an active thromboembolic event (within the last 24 hours) i.e. active stroke, myocardial infarction, or pulmonary embolism
* Any patient with a hypersensitivity or anaphylactic reaction to TXA
* Any patient more than 3 hours post injury
* Traumatic arrest with > 5 minutes CPR without return of vital signs
* Penetrating cranial injury
* Traumatic brain injury with brain matter exposed
* Isolated drowning or hanging victims
* Documented cervical cord injury with motor deficit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Survival at 24 hours | 24 hours
  Mortality at 24 hours
Survival at 48 hours | 48 hours
  Mortality at 48 hours
Survival at 28 days | 28 days
  Mortality at 28 days

SECONDARY OUTCOMES:
Blood Transfusion | 24 hours
  Units of blood products needed (<2 units, 2-4 units, >4 units)
Length of Hospital Stay | 28 days
  Duration of ICU stay
Adverse Events | 28 days
  Incidence of known adverse events associated with TXA

CONTACTS AND LOCATIONS:
Overall Officials: Michael Neeki, Principal Investigator — Arrowhead Regional Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CRASH-2 collaborators; Roberts I, Shakur H, Afolabi A, Brohi K, Coats T, Dewan Y, Gando S, Guyatt G, Hunt BJ, Morales C, Perel P, Prieto-Merino D, Woolley T. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomised controlled trial. Lancet. 2011 Mar 26;377(9771):1096-101, 1101.e1-2. doi: 10.1016/S0140-6736(11)60278-X. PMID 21439633
- [Background] Morrison JJ, Dubose JJ, Rasmussen TE, Midwinter MJ. Military Application of Tranexamic Acid in Trauma Emergency Resuscitation (MATTERs) Study. Arch Surg. 2012 Feb;147(2):113-9. doi: 10.1001/archsurg.2011.287. Epub 2011 Oct 17. PMID 22006852
- [Result] Neeki MM, Dong F, Toy J, Vaezazizi R, Powell J, Jabourian N, Jabourian A, Wong D, Vara R, Seiler K, Pennington TW, Powell J, Yoshida-McMath C, Kissel S, Schulz-Costello K, Mistry J, Surrusco MS, O'Bosky KR, Van Stralen D, Ludi D, Sporer K, Benson P, Kwong E, Pitts R, Culhane JT, Borger R. Efficacy and Safety of Tranexamic Acid in Prehospital Traumatic Hemorrhagic Shock: Outcomes of the Cal-PAT Study. West J Emerg Med. 2017 Jun;18(4):673-683. doi: 10.5811/westjem.2017.2.32044. Epub 2017 Apr 19. PMID 28611888

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT03469947/Prot_SAP_000.pdf